CLINICAL TRIAL: NCT04153136
Title: Ending Subclinical Heart Failure Using an Aldosterone and Natriuretic Peptide Targeted Treatment in HIV--The ENCHANTMENT HIV Study
Brief Title: The ENCHANTMENT HIV Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Suman Srinivasa, M.D., Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MGH2019P002355
Record Dates: First submitted 2019-10-30; First posted 2019-11-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: HIV/AIDS; Heart Failure With Preserved Ejection Fraction
Keywords: HIV; Sacubitril/valsartan; Heart Failure with Preserved Ejection Fraction; Aldosterone; Natriuretic Peptides; Myocardial Dysfunction; Cardiovascular Disease
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cardiovascular Diseases | interventions — sacubitril and valsartan sodium hydrate drug combination; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacubitril/Valsartan (Experimental): Sacubitril/Valsartan 49-51mg twice daily along with lifestyle modification (counseling regarding diet and healthy activity) for 6 months
  Interventions: Drug: Sacubitril-Valsartan 49-51Mg Oral Tablet
- Placebo (Placebo Comparator): Placebo twice daily along with lifestyle modification (counseling regarding diet and healthy activity) for 6 months
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Sacubitril-Valsartan 49-51Mg Oral Tablet — By mouth twice daily
  Other Names: Entresto
  Arms: Sacubitril/Valsartan
Drug: Placebo oral tablet — Placebo oral tablet By mouth twice daily
  Arms: Placebo

SUMMARY:
Persons with HIV, even those well-treated, are at increased risk for heart disease when compared to the general population. Two hormones called aldosterone and brain natriuretic peptide (BNP), which have been shown to be abnormal in HIV, may be associated with inflammation as well as early changes in structure and function of the heart. This study is being conducted to evaluate whether therapies to block aldosterone and increase BNP levels may reduce the burden and progression of heart failure to improve cardiovascular health.

DETAILED DESCRIPTION:
This is a 6-month study enrolling persons with HIV with no known history of heart disease. Participants will be screened for early signs of heart failure using cardiac ultrasound (cardiac transthoracic echocardiography or cardiac TTE). Those participants who have early changes in the structure and function of the heart and may be at future risk for heart failure will be enrolled into the study. Additional imaging of the heart will occur using cardiac magnetic resonance imaging (cardiac MRI). Following baseline studies, participants will either receive a medication called sacubitril/valsartan or placebo for 6 months. Sacubitril/valsartan in an FDA approved medication currently being used for heart failure with reduced ejection fraction in the general population, and we are evaluating whether this medication could be useful to reduce HIV-related heart failure with preserved ejection fraction. Sacubitril/valsartan is an oral medication taken twice daily that may block aldosterone hormone and increase natriuretic peptide hormone. Overall, this study aims to investigate the effect of sacubitril/valsartan on measures of heart disease related to inflammation, structure and function of the heart muscle in HIV using cardiac TTE and cardiac MRI imaging as well as blood markers of heart failure and inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Antiretroviral therapy use for >12 months
2. HIV Viral Load <200 copies/mL
3. Left Ventricular Ejection Fraction>50%
4. Demonstration of one or more criteria for myocardial dysfunction on cardiac transthoracic echocardiogram, relevant to the progression of heart failure with preserved ejection fraction:

   * Left Atrial Volume Index > 28 mL/m2
   * Global Longitudinal Strain <18%
   * Left Ventricular Mass Index > 95g/m2 (female), 115 g/m2 (male)

Exclusion Criteria:

1. Known history of congestive heart failure or valvular disease
2. Recent cardiac event or stroke within 3 months
3. Current medication use acting along the RAAS pathway (ACEi, ARB, MR blockade, direct renin inhibitor), potassium (K) supplementation or diuretic
4. Angioedema to ACEi or ARB
5. SBP<100 mmHg
6. Medication suspected to have contraindication with active study drug
7. Steroid use within last 3 months
8. Uncontrolled diabetes requiring insulin and/or HbA1c > 7.5%
9. Creatinine (Cr)>1.5 mg/dL and estimated GFR<60 mL/min/1.73m2
10. K>5.5 mEq/L
11. Hemoglobin <10.0 g/dL
12. Known liver disease or ALT>3x upper limit normal
13. Pregnant, actively seeking pregnancy or breastfeeding
14. Estrogen, progestin derivative, or other sex steroid use within 3 months. Stable physiologic testosterone replacement (> 3 months) is acceptable
15. Current bacterial or other infection
16. Active substance abuse
17. Known reaction to gadolinium

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Myocardial Inflammation/Fibrosis | 6 months
  Myocardial Inflammation/Fibrosis measured by extracellular volume fraction via cardiac magnetic resonance imaging
Myocardial Dysfunction | 6 months
  Left Atrial Volume Index or Global Longitudinal Strain measured by cardiac transthoracic echocardiography

SECONDARY OUTCOMES:
Other Indices of Myocardial Dysfunction | 6 months
  Alterations in other cardiac structure and function as measured by cardiac magnetic resonance imaging or cardiac transthoracic echocardiogram
Markers of Myocardial Inflammation and Fibrosis | 6 months
  Circulating biomarkers of myocardial inflammation and fibrosis: Gal3, ST2, GDF15, hs-cTnT
Cardiac Natriuretic Peptides | 6 months
  Circulating cardiac natriuretic peptides: ANP, BNP, NT-proBNP

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srinivasa S, Fitch KV, Wong K, Torriani M, Mayhew C, Stanley T, Lo J, Adler GK, Grinspoon SK. RAAS Activation Is Associated With Visceral Adiposity and Insulin Resistance Among HIV-infected Patients. J Clin Endocrinol Metab. 2015 Aug;100(8):2873-82. doi: 10.1210/jc.2015-1461. Epub 2015 Jun 18. PMID 26086328
- [Background] Murphy CA, Fitch KV, Feldpausch M, Maehler P, Wong K, Torriani M, Adler GK, Grinspoon SK, Srinivasa S. Excessive Adiposity and Metabolic Dysfunction Relate to Reduced Natriuretic Peptide During RAAS Activation in HIV. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1558-1565. doi: 10.1210/jc.2017-02198. PMID 29408981
- [Background] Srinivasa S, Fitch KV, Wong K, O'Malley TK, Maehler P, Branch KL, Looby SE, Burdo TH, Martinez-Salazar EL, Torriani M, Lyons SH, Weiss J, Feldpausch M, Stanley TL, Adler GK, Grinspoon SK. Randomized, Placebo-Controlled Trial to Evaluate Effects of Eplerenone on Metabolic and Inflammatory Indices in HIV. J Clin Endocrinol Metab. 2018 Jun 1;103(6):2376-2384. doi: 10.1210/jc.2018-00330. PMID 29659888

DOCUMENTS (1):
  • Informed Consent Form (2025-08-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT04153136/ICF_000.pdf